CLINICAL TRIAL: NCT02630316
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Inhaled Treprostinil in Subjects With Pulmonary Hypertension Due to Parenchymal Lung Disease
Brief Title: Safety and Efficacy of Inhaled Treprostinil in Adult PH With ILD Including CPFE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PH-201
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease; Combined Pulmonary Fibrosis and Emphysema
Keywords: Treprostinil; PH; ILD; CPFE; 6 Minute Walk Test
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Emphysema | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo inhaled using an ultrasonic nebulizer four times daily
  Interventions: Drug: Placebo
- Inhaled Treprostinil (Active Comparator): Active Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled four times daily and titrated up to a maximum of 12 breaths four times daily
  Interventions: Drug: Inhaled Treprostinil

INTERVENTIONS:
Drug: Inhaled Treprostinil — Inhaled treprostinil (6 mcg/breath) administered four times daily
  Other Names: Tyvaso
  Arms: Inhaled Treprostinil
Drug: Placebo — Placebo administered four times daily
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized (1:1 inhaled treprostinil: placebo), double-blinded, placebo-controlled trial to evaluate the safety and efficacy of inhaled treprostinil in subjects with pre-capillary pulmonary hypertension (PH) associated with interstitial lung disease (ILD) including combined pulmonary fibrosis and emphysema (CPFE). The study included 326 patients at approximately 120 clinical trial centers. The treatment phase of the study lasted approximately 16 weeks. Patients who completed all required assessments were eligible to enter an open-label, extension study (RIN-PH-202).

DETAILED DESCRIPTION:
Study RIN-PH-201 was a multicenter, randomized, double-blind, placebo controlled, 16 week, parallel group study designed to investigate the safety and efficacy of inhaled treprostinil in subjects with PH-ILD. Subjects initiated inhaled treprostinil or placebo at a dose of 3 breaths (18 mcg) 4 times daily (QID) (during waking hours). Study drug doses were maximized throughout the study. Dose escalations (additional 1 breath QID) could occur up to every 3 days with a target dosing regimen of 9 breaths (54 mcg) QID and a maximum dose of 12 breaths (72 mcg) QID, as clinically tolerated. Subjects were assessed during Screening and Baseline to determine eligibility for the study. Once eligible, 5 Treatment Phase visits to the clinic were required at Week 4, Week 8, Week 12, Week 15, and Week 16 (final study visit). An Early Termination (ET) Visit was conducted for subjects who discontinued prior to Week 16; all assessments planned for the final Week 16 Visit were conducted during the ET Visit, if applicable. Subjects were contacted at least weekly by telephone or email to assess tolerance to study drug, AEs, and changes to concomitant medications. Efficacy assessments consisted of 6-minute walk distance (6MWD), plasma N-terminal prohormone brain natriuretic peptide (NT-proBNP) concentration, and incidence of clinical worsening. Exploratory endpoints included change in St. George's Respiratory Questionnaire (SGRQ), change in distance saturation product (DSP), time to exacerbation of underlying lung disease, and pulmonary function tests (PFT). Safety assessments consisted of the development of AEs, vital signs, clinical laboratory parameters, ECG parameters, hospitalizations due to cardiopulmonary indications, exacerbations of underlying lung disease, and oxygenation. Subjects who remained on study drug, completed all assessments during the 16-week Treatment Phase, and met all eligibility criteria were eligible for the open-label extension study (RIN-PH-202). Additionally, subjects who withdrew from study drug prior to Week 16 due to clinical worsening and returned to the clinic for scheduled visits (excluding the Week 15 Visit) were eligible for RIN PH-202.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily gave informed consent to participate in the study.
2. Males and females aged 18 years or older at the time of informed consent.

   a. Females of reproductive potential were non-pregnant (as confirmed by a urine pregnancy test at screening) and non-lactating, and: i. Abstained from intercourse (when in line with their preferred and usual lifestyle), or ii. Used 2 medically acceptable, highly effective forms of contraception for the duration of study, and at least 30 days after discontinuing study drug.

   b. Males with a partner of childbearing potential used condoms for the duration of treatment and for at least 48 hours after discontinuing study drug.
3. The subject had a confirmed diagnosis of WHO Group 3 PH based on computed tomography (CT) imaging which was performed within 6 months prior to randomization and demonstrated evidence of diffuse parenchymal lung disease. Subjects had any form of ILD or CPFE.
4. Subjects were required to have a right heart catheterization (RHC) within 1 year prior to randomization with the following documented parameters:

   1. Pulmonary vascular resistance (PVR) >3 Wood Units (WU) and
   2. A pulmonary capillary wedge pressure (PCWP) of <15 mmHg and
   3. A mean pulmonary arterial pressure (mPAP) of >25 mmHg
5. Baseline 6MWD ≥100 m.
6. Subjects on a chronic medication for underlying lung disease (ie, pirfenidone, nintedanib, etc) were on a stable and optimized dose for ≥30 days prior to randomization.
7. In the opinion of the Investigator, the subject was able to communicate effectively with study personnel, and was considered reliable, willing and likely to be cooperative with protocol requirements, including attending all study visits.
8. Subjects with connective tissue disease (CTD) had a Baseline forced vital capacity (FVC) of <70%.

Exclusion criteria:

1. The subject had a diagnosis of PAH or PH for reasons other than WHO Group 3 PH ILD as outlined in Inclusion Criterion 3.
2. The subject showed intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to effectively titrate that therapy.
3. The subject received any PAH-approved therapy including: prostacyclin therapy (ie, epoprostenol, treprostinil, iloprost, or beraprost; except for acute vasoreactivity testing), prostacyclin (IP) receptor agonist (selexipag), endothelin receptor antagonist (ERA), phosphodiesterase type 5 inhibitor (PDE5-I), or soluble guanylate cyclase (sGC) stimulator within 60 days of randomization.
4. The subject had evidence of clinically significant left-sided heart disease as defined by:

   1. PCWP >15 mmHg
   2. Left ventricular ejection fraction <40%. Note: Subjects with abnormal left ventricular function attributable entirely to impaired left ventricular filling due to the effects of right ventricular overload (ie, right ventricular hypertrophy and/or dilatation) were not excluded.
5. The subject was receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
6. Current use of any inhaled tobacco/marijuana products or significant history of drug abuse at the time of informed consent.
7. Exacerbation of underlying lung disease or active pulmonary or upper respiratory infection within 30 days of randomization.
8. Initiation of pulmonary rehabilitation within 12 weeks prior to randomization.
9. In the opinion of the Investigator, the subject had any condition that would interfere with the interpretation of study assessments or has any disease or condition (ie, peripheral vascular disease, musculoskeletal disorder, morbid obesity) that would likely be the primary limit to ambulation (as opposed to PH).
10. Use of any investigational drug/device, or participation in any investigational study with therapeutic intent within 30 days prior to randomization.
11. Severe concomitant illness limiting life expectancy (<6 months).
12. Acute pulmonary embolism within 90 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (96):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - IMC-Diagnostic & Medical Clinic, Mobile, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Advanced Health Sciences Pavilion, Beverly Hills, California
  - University of California San Francisco - Fresno, Fresno, California
  - University of California San Diego, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - University of Southern California Health Sciences, Los Angeles, California
  - Department of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Pacific Pulmonary Medical Group, Riverside, California
  - Kaiser Permanente - Roseville, Roseville, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente, San Francisco, California
  - University of Colorado Hospital - Cardiac and Vascular Center, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Lung, Asthma & Sleep Specialists, P.A., Celebration, Florida
  - St. Francis Sleep, Allergy and Lung Institute, Clearwater, Florida
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - St. Vincent's Health System, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - South Miami Heart Specialists, South Miami, Florida
  - Tampa General Hospital Center of Research Excellence, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Piedmont - Georgia Lung Associates, Austell, Georgia
  - Wellstar Medical Group - Pulmonary Medicine, Marietta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - U Health Physicians Advanced Heart and Lung Clinic, Indianapolis, Indiana
  - Community Heart and Vascular Hospital East, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - Louisiana State University Health Sciences Center New Orleans, New Orleans, Louisiana
  - Chest Medicine Associates, South Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Pulmonary and Critical Care Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Spectrum Health Heart and Lung Specialized Care Clinic, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Northwell Health, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian - Weill Cornell Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center-Duke South Clinic, Durham, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Health, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Montifiore University Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Statcare Pulmonary Consultants, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Houston Methodist, Houston, Texas
  - Memoral Hermann Hospital - Texas Medical Center, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Vermont Lung Center, Colchester, Vermont
  - Inova Fairfax Medical Campus, Fairfax, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Auxilio Mutuo Hospital, Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Nathan SD, Deng C, King CS, DuBrock HM, Elwing J, Rajagopal S, Rischard F, Sahay S, Broderick M, Shen E, Smith P, Tapson VF, Waxman AB. Inhaled Treprostinil Dosage in Pulmonary Hypertension Associated With Interstitial Lung Disease and Its Effects on Clinical Outcomes. Chest. 2023 Feb;163(2):398-406. doi: 10.1016/j.chest.2022.09.007. Epub 2022 Sep 15. PMID 36115497
- [Derived] Nathan SD, Waxman A, Rajagopal S, Case A, Johri S, DuBrock H, De La Zerda DJ, Sahay S, King C, Melendres-Groves L, Smith P, Shen E, Edwards LD, Nelsen A, Tapson VF. Inhaled treprostinil and forced vital capacity in patients with interstitial lung disease and associated pulmonary hypertension: a post-hoc analysis of the INCREASE study. Lancet Respir Med. 2021 Nov;9(11):1266-1274. doi: 10.1016/S2213-2600(21)00165-X. Epub 2021 Jun 29. PMID 34214475
- [Derived] Waxman A, Restrepo-Jaramillo R, Thenappan T, Ravichandran A, Engel P, Bajwa A, Allen R, Feldman J, Argula R, Smith P, Rollins K, Deng C, Peterson L, Bell H, Tapson V, Nathan SD. Inhaled Treprostinil in Pulmonary Hypertension Due to Interstitial Lung Disease. N Engl J Med. 2021 Jan 28;384(4):325-334. doi: 10.1056/NEJMoa2008470. Epub 2021 Jan 13. PMID 33440084

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Inhaled Treprostinil
Started | 163 | 163
Completed | 128 | 130
Not Completed | 35 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Inhaled Treprostinil | Total
Number analyzed (Participants) | 163 | 163 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 64 | 112
  >=65 years | 115 | 99 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.2) | 65.6 (12.7) | 66.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 85 | 153
  Male | 95 | 78 | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 41 | 71
  White | 126 | 112 | 238
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2 | 0 | 2
  United States | 161 | 163 | 324
Weight [Mean (Standard Deviation); unit: kg] | 83.5 (20.6) | 83.9 (20.5) | 83.7 (20.5)
Height [Mean (Standard Deviation); unit: cm] — Population: Height was not collected for 1 subject in the Placebo group and 1 subject in the Inhaled Treprostinil group.
  cm
    number analyzed (Participants) | 162 | 162 | 324
    (all) | 169.0 (9.4) | 167.5 (10.3) | 168.2 (9.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Height was not collected for 1 subject in the Placebo group and 1 subject in the Inhaled Treprostinil group.
  kg/m^2
    number analyzed (Participants) | 162 | 162 | 324
    (all) | 29.0 (5.9) | 30.0 (6.6) | 29.5 (6.3)
6 Minute Walk Distance [Mean (Standard Deviation); unit: meters] | 265.1 (93.1) | 254.1 (102.4) | 259.6 (97.9)
N-terminal prohormone brain natriuretic peptide (NT-proBNP) [Mean (Standard Deviation); unit: pg/mL] — Population: NT-proBNP was not collected for 10 subjects from the Inhaled Treprostinil group and 5 subjects from the Placebo group.
  pg/mL
    number analyzed (Participants) | 158 | 153 | 311
    (all) | 210.9 (370.7) | 223.5 (378.5) | 217.1 (374.0)
Pulmonary Vascular Resistance (PVR) [Mean (Standard Deviation); unit: Wood Units (WU)] | 6.0 (2.7) | 6.4 (2.9) | 6.2 (2.8)
Mean pulmonary arterial pressure (PAPm) [Mean (Standard Deviation); unit: mmHg] | 36.0 (8.4) | 37.2 (8.6) | 36.6 (8.5)
Pulmonary Capillary Wedge Pressure (PCWP) [Mean (Standard Deviation); unit: mmHg] | 9.6 (3.5) | 10.1 (3.4) | 9.8 (3.5)
Vasodilator testing during confirmatory right heart catheterization (RHC)? [Count of Participants; unit: Participants]
  Yes | 45 | 42 | 87
  No | 118 | 121 | 239
10 mmHg decrease in PAPm during Confirmatory RHC? [Count of Participants; unit: Participants]
  Yes | 8 | 6 | 14
  No | 35 | 37 | 72
  Not tested | 120 | 120 | 240
Vasodilator medications used during Confirmatory RHC? [Count of Participants; unit: Participants]
  Inhaled Nitrous Oxide | 43 | 39 | 82
  Adenosine | 2 | 1 | 3
  Other | 0 | 2 | 2
  No medication | 118 | 121 | 239

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Distance (6MWD) Measured at Peak Exposure From Baseline to Week 16
Description: The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Week 16, correlates with the current clinical standard for assessing patient functional status in the treatment of PH and is considered an objective measure of patient functional status. Subjects will be instructed to walk down a corridor at a comfortable speed as far as they can manage for six minutes. Peak exposure 6MWD will occur by conducting 6-minute walk test (6MWT) within 10 to 60 minutes after the most recent dose of study drug dose.
Time Frame: Baseline and Week 16
Population: All Subjects Dosed
Measure: Median (Full Range); unit: meters
Arm/Group | Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 163 | 163
meters | -9.0 [-426 to 179] | 6.0 [-396 to 183]
Statistical Analysis 1: Comparison: Placebo vs Inhaled Treprostinil; Test type: Superiority; p = 0.0043, ANCOVA — p-value is obtained from nonparametric ANCOVA adjusted for Baseline 6MWD category; Hodges-Lehmann = 21.0, 95% CI 2-sided [7.0 to 37.0]

2. Secondary Outcome: Change in Plasma Concentration of N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) From Baseline to Week 16
Description: The NT-proBNP serum concentration is a useful biomarker associated with changes in right heart morphology and function. NT-proBNP serum concentration will be assessed to compare the severity of heart failure at Baseline and Week 16. Blood for NT-proBNP assessment must be drawn prior to conducting the 6MWT.
Time Frame: Baseline and Week 16
Population: Only subjects with Baseline NT-proBNP are included. For subjects who do not have Week 16 measure, the last observation carried forward imputation is used.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 160 | 156
pg/mL | 20.65 [-5483.3 to 87148.3] | -22.65 [-11433.0 to 5373.1]
Statistical Analysis 1: Comparison: Placebo vs Inhaled Treprostinil; Test type: Superiority; p < 0.0001, ANCOVA

3. Secondary Outcome: Incidence of Clinical Worsening
Description: Subjects were monitored for clinical worsening from the time of randomization until 1 of the following criteria were met: hospitalization due to a cardiopulmonary indication; decrease in 6MWD >15% from Baseline directly related to the disease under study, at 2 consecutive visits and at least 24 hours apart; death (all causes); or lung transplantation.
Time Frame: Baseline to Week 16
Population: All Subjects with Clinical Worsening Events
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 163 | 163
Participants | 54 | 37
Statistical Analysis 1: Comparison: Placebo vs Inhaled Treprostinil; Test type: Superiority; p = 0.0410, Log Rank — p-value is calculated with log-rank test stratified by baseline 6MWD category; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.40 to 0.92] — p-value was 0.0202 for the proportional hazard model. Hazard ratio, 95% confidence interval (CI), and p-values are calculated with proportional hazards model with treatment and Baseline 6MWD (continuous) as explanatory variables

4. Secondary Outcome: Change in Peak 6-minute Walk Distance (6MWD) From Baseline to Week 12
Description: The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Week 12, correlates with the current clinical standard for assessing patient functional status in the treatment of PH and is considered an objective measure of patient functional status. Subjects will be instructed to walk down a corridor at a comfortable speed as far as they can manage for six minutes. Peak exposure 6MWD will occur by conducting 6MWT within 10 to 60 minutes after the most recent dose of study drug dose.
Time Frame: Baseline and Week 12
Population: For those subjects who withdrew early due to death, were too ill to walk, or had no 6MWD measure due to clinical worsening event, the 6MWD is set to 0, for all other withdrawals without Week 12 measurement, last observation carried forward (LOCF) is used for imputation.
Measure: Median (Full Range); unit: meters
Arm/Group | Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 163 | 163
meters | -3.0 [-369 to 152] | 8.0 [-360 to 192]
Statistical Analysis 1: Comparison: Placebo vs Inhaled Treprostinil; Test type: Superiority; p = 0.0041, ANCOVA — p-value is obtained from nonparametric ANCOVA adjusted for Baseline 6MWD category; Hodges-Lehmann = 20.0, 95% CI 2-sided [7.0 to 34.0]

5. Secondary Outcome: Change in Trough 6-minute Walk Distance (6MWD) From Baseline to Week 15
Description: The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Week 15, correlates with the current clinical standard for assessing patient functional status in the treatment of PH and is considered an objective measure of patient functional status. Subjects will be instructed to walk down a corridor at a comfortable speed as far as they can manage for six minutes. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation. Trough exposure 6MWD will occur by conducting 6-minute walk test (6MWT) at least four hours after the most recent study drug dose.
Time Frame: Baseline and Week 15
Population: For those subjects who withdrew early due to death, were too ill to walk, or had no 6MWD measure due to clinical worsening event, the 6MWD is set to 0, for all other withdrawals without Week 15 measurement, baseline observation carried forward is used for imputation.
Measure: Median (Full Range); unit: meter
Arm/Group | Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 163 | 163
meter | -9.0 [-369 to 180] | 0.0 [-396 to 144]
Statistical Analysis 1: Comparison: Placebo vs Inhaled Treprostinil; Test type: Superiority; p = 0.0432, ANCOVA — p-value is obtained from nonparametric ANCOVA adjusted for Baseline 6MWD category; Hodges-Lehmann = 15.0, 95% CI 2-sided [0.0 to 29.0]

ADVERSE EVENTS:
Time Frame: AEs were recorded throughout the course of the study from the time that each subject signed the ICF until all study assessments were completed (16 weeks).
Description: All AEs were followed until either resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, or for at least 30 days if the AE extended beyond the final study visit. All AEs which met the criteria for serious (ie, SAEs) were followed until resolution, death, or the subject was lost to follow-up even if they were ongoing more than 30 days after completion of the final study visit (Week 16 or early termination Visit).
Groups:
- Active Inhaled Treprostinil: Active Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled four times daily and titrated up to a maximum of 12 breaths four times daily
  Inhaled Treprostinil: Inhaled treprostinil (6 mcg/breath) administered four times daily
Arm/Group | Placebo | Active Inhaled Treprostinil
All-Cause Mortality (participants affected / at risk) | 12/163 | 10/163
Serious Adverse Events (participants affected / at risk) | 42/163 | 38/163
Other Adverse Events (participants affected / at risk) | 149/163 | 152/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=163) | Active Inhaled Treprostinil (N=163)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (2)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Chronic right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9) | 1 (1)
Rhinovirus infetion (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (11) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=163) | Active Inhaled Treprostinil (N=163)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (56) | 71 (76)
Headache (Nervous system disorders) | 32 (34) | 45 (49)
Nausea (Gastrointestinal disorders) | 26 (27) | 25 (26)
Diarrhea (Gastrointestinal disorders) | 19 (19) | 22 (24)
Fatigue (General disorders) | 23 (24) | 23 (24)
Chest pain (General disorders) | 5 (5) | 14 (14)
Oedema peripheral (General disorders) | 10 (11) | 13 (13)
Chest discomfort (General disorders) | 4 (4) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 11 (12)
Pneumonia (Infections and infestations) | 11 (12) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 8 (8)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 25 (25) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 7 (7)
Dizziness (Nervous system disorders) | 23 (23) | 30 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 (56) | 41 (46)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 20 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 18 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02630316/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT02630316/SAP_003.pdf